CLINICAL TRIAL: NCT02362893
Title: Treatment of Hypertension: an Interventional Approach to Improve Blood Pressure Control
Acronym: DRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ulla Hjørnholm, RN MSc, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/159
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hypertension
Keywords: Hypertension; Adherence; Direct Observed Therapy (DOT); RCT
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Direct Observed Therapy (Experimental): Direct Observed Therapy immediately followed by mounting of ambulatory blood pressure device and measurement of ambulatory blood pressure according to ESH 2013 guidelines.
  Interventions: Other: Direct Observed Therapy
- Control (No Intervention): Standard care

INTERVENTIONS:
Other: Direct Observed Therapy — Patients allocated to the intervention group take their medication (from original blister packaged) in front of the invistigator who observe the patient swallowing the medication. To secure the principals of Direct Observed Therapy, the patient do not leave the clinic for two hours.
  Other Names: DOT
  Arms: Direct Observed Therapy

SUMMARY:
The purpose of the study is to access the change in mean daytime systolic blood pressure in participants with essential hypertension not adequately controlled (defined as mean systolic daytime ambulatory blood pressure ≥ 135 mmHg) and randomly assigned to either an intervention group with one-time only Direct Observed Therapy (DOT) immediately followed by ABPM or a control group with standard ABPM.

DETAILED DESCRIPTION:
More than 1 billion people world wide suffer from hypertension (HT), leaving it the world´s top rank risk factor and contributor to global disease burden. Cardiac disease, stroke, kidney disease and dementia are diseases related to HT with high economic burden on societies and each year 9.4 million people die as a direct consequence of HT.

Estimated < 50 % of hypertensive patients adhere to preventive hypertensive medication after 1 year of treatment.

Poor adherence to antihypertensive treatment have by many been explained partly by the silent nature of hypertension, the risk of side effects from antihypertensive medication, treatment expenditures and the patient health perspectives.

In a randomized controlled trial design we plan to enrol 20 subjects, the limited number explained by the study being part of the initial planning of a larger scale trial organized by the research group, to invistigate the change in ambulatory bloodpressure with or with out Direct Observed Theraphy prior to meassurement, as a one-time-only medication adherence check.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Residing in Oslo/Akershus
* Ambulatory Systolic Daytime Blood Pressure ≥ 135 mmHg
* ≥ 2 antihypertensive medications
* Be able to read and write Norwegian

Exclusion Criteria:

* Critical illness, ongoing treatment
* Known atrial fibrillation
* Known heart valve stenosis
* Myocardial infarction, angina pectoris or stroke the past 6 months
* Known severe renal impairment (eGFR < 30 ml/min/1.73 m2)
* History of DOT prior to ABPM
* Participation in other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2018-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory mean systolic daytime blood pressure | Measurement at follow-up visit 3 weeks ± 7 days relative to baseline.

SECONDARY OUTCOMES:
Change in mean office systolic blood pressure | Measurement at follow-up visit 3 weeks ± 7 days relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Aud Høieggen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fadl Elmula FE, Hoffmann P, Fossum E, Brekke M, Gjonnaess E, Hjornholm U, Kjaer VN, Rostrup M, Kjeldsen SE, Os I, Stenehjem AE, Hoieggen A. Renal sympathetic denervation in patients with treatment-resistant hypertension after witnessed intake of medication before qualifying ambulatory blood pressure. Hypertension. 2013 Sep;62(3):526-32. doi: 10.1161/HYPERTENSIONAHA.113.01452. Epub 2013 Jul 8. PMID 23836798
- [Background] Fadl Elmula FE, Hoffmann P, Larstorp AC, Fossum E, Brekke M, Kjeldsen SE, Gjonnaess E, Hjornholm U, Kjaer VN, Rostrup M, Os I, Stenehjem A, Hoieggen A. Adjusted drug treatment is superior to renal sympathetic denervation in patients with true treatment-resistant hypertension. Hypertension. 2014 May;63(5):991-9. doi: 10.1161/HYPERTENSIONAHA.114.03246. Epub 2014 Mar 3. PMID 24591332